CLINICAL TRIAL: NCT00165360
Title: A Phase II Study of Prolonged Daily Temozolomide for Low-Grade Glioma
Brief Title: Prolonged Daily Temozolomide for Low-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Schering-Plough (Industry); Brigham and Women's Hospital (Other); University of Virginia (Other)
Responsible Party: Patrick Wen, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-111
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Glioma; Astrocytoma; Oligodendroglioma
Keywords: low-grade glioma; astrocytoma; oligodendroglioma; oligoastrocytoma; temozolomide; mixed oligoastrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Temozolomide — Given once daily for 49 days followed by 28 days with no drug for a maximum of a year and a half

SUMMARY:
The purpose of this trial is to determine the effects (good and bad) temozolomide has on patients with low-grade glioma. It will also determine whether temozolomide is effective in preventing or delaying future tumor growth.

DETAILED DESCRIPTION:
* Treatment with temozolomide is based upon an 11-week cycle (7 weeks on the drug and 4 weeks off). Patients will receive temozolomide once daily for 49 days, then have 28 days without taking temozolomide.
* Every two to four weeks a physical and neurological examination and blood work will be performed. A magnetic resonance imaging (MRI) scan of the patient's brain will be done approximately every three months (before each cycle of treatment).
* Treatment may continue for a maximum of a year and a half based on 6 eleven-week cycles. The actual duration of therapy will depend upon the response to treatment and the development of side effects or toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of a low-grade glioma (astrocytoma, oligodendroglioma, or mixed oligoastrocytoma)
* Measurable disease on MRI
* Patients that have undergone recent resection for newly diagnosed or recurrent or progressive tumor are eligible if they have recovered from the effects of surgery.
* Patients with recurrent disease my have had one prior chemotherapy regimen
* Older than 18 years of age.
* Karnofsky performance status (KPS) performance score of > 70%
* Adequate hematologic, renal and liver functions,
* Life expectancy of greater than 12 weeks.
* Negative pregnancy test.

Exclusion Criteria:

* Prior treatment with temozolomide
* Patients who are not neurologically stable
* Acute infection treated with intravenous antibiotics
* Non-malignant systemic disease
* Frequent vomiting, inability to swallow or a medical condition that could interfere with oral medication.
* Previous or concurrent malignancies at other sites, with the exception of surgically cured carcinoma in-situ of the cervix, and basal or squamous cell carcinoma of the skin.
* HIV positive or AIDS-related illness
* Pregnant or nursing women
* Patients with allergy to decarbazine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2001-09; Primary Completion 2006-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine the effects temozolomide has on low-grade gliomas | 3 years

SECONDARY OUTCOMES:
To determine whether temozolomide is effective in preventing or delaying future tumor growth | 3 years
to determine the safety of temozolomide | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts